CLINICAL TRIAL: NCT01894737
Title: The Effect of Creatine Supplementation on Muscle Loss During Immobilisation
Brief Title: The Effect of Creatine on Muscle Loss
Acronym: CML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 13-3-023
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Muscle Loss
MeSH Terms: conditions — Muscular Atrophy | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- immobilisation and placebo (Placebo Comparator): Seven days of one-legged knee immobilisation with placebo supplementation
  Interventions: Other: Placebo supplementation
- immobilisation and creatine (Experimental): Seven days of one-legged knee immobilisation with creatine supplementation
  Interventions: Other: Creatine supplementation

INTERVENTIONS:
Other: Placebo supplementation — Seven days of one-legged knee immobilisation with placebo supplementation
  Arms: immobilisation and placebo
Other: Creatine supplementation — Seven days of one-legged knee immobilisation with creatine supplementation.
  Arms: immobilisation and creatine

SUMMARY:
The primary aim of this study is to determine the effect of creatine supplementation on muscle mass loss during short-term immobilisation in healthy, young people.

DETAILED DESCRIPTION:
Seven days of one-legged knee immobilisation in young subjects with creatine or Placebo supplementation. A randomly selected leg is immobilized for seven days. Muscle mass and strength will be determined and muscle biopsies will be collected before and immediately after immobilisation. A week after the cast is removed we will assess any differences in recovery between intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged from 18-35 years
* 18.5 < BMI < 30 kg/m2

Exclusion Criteria:

* (Family) history of thrombosis
* Smoking
* Recent surgery
* Performing regular resistance training more than once per week in the past year
* Any back/leg/knee/shoulder complaints which may interfere with the use of crutches
* Current systemic use of corticosteroids, growth hormone, testosterone, immunosuppressants or insulin
* All co-morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. arthritis, spasticity/rigidity, all neurological disorders and paralysis)
* Use of anti-coagulants
* Pre-existing renal disease or those with a potential risk for renal dysfunction (diabetes, hypertension, reduced glomerular filtration rate)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
change in quadriceps muscle cross-sectional area (CSA) | Before and after 1 week of immobilisation, and after 1 week of recovery
  immediately before and after 1 week of immobilisation, and after 1 week recovery, quadriceps CSA will be assessed

SECONDARY OUTCOMES:
change in muscle fiber type specific CSA | Before and after 1 week of immobilisation, and after 1 week of recovery
  immediately before and after 1 week of immobilization, and after 1 week of natural recovery
change in muscle strength | before and after 1 week of immobilisation, and after 1 week of recovery
  immediately before and after 1 week of immobilization, and after 1 week of natural recovery, one-repetition maximum (1RM) muscle strength will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Backx EMP, Hangelbroek R, Snijders T, Verscheijden ML, Verdijk LB, de Groot LCPGM, van Loon LJC. Creatine Loading Does Not Preserve Muscle Mass or Strength During Leg Immobilization in Healthy, Young Males: A Randomized Controlled Trial. Sports Med. 2017 Aug;47(8):1661-1671. doi: 10.1007/s40279-016-0670-2. PMID 28054322
- [Derived] Dirks ML, Backx EM, Wall BT, Verdijk LB, van Loon LJ. May bed rest cause greater muscle loss than limb immobilization? Acta Physiol (Oxf). 2016 Sep;218(1):10-2. doi: 10.1111/apha.12699. Epub 2016 May 20. No abstract available. PMID 27124248